CLINICAL TRIAL: NCT03929068
Title: Sinemet in ALS and PLS
Brief Title: Sinemet for Spasticity and Function in Amyotrophic Lateral Sclerosis and Primary Lateral Sclerosis
Acronym: ALS and PLS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Sinemet-001
Record Dates: First submitted 2019-04-10; First posted 2019-04-26 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
Keywords: ALS; PLS; Primary Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Intervention Model Description: Identified participants will be randomized to receive either placebo or carbidopa-levodopa for a period of three weeks before crossing over to the other arm of the study. The two periods will be separated by a one day washout period.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- carbidopa-levodopa (Active Comparator): Each tablet of carbidopa-levodopa in this study will be equivalent to half of a standard carbidopa-levodopa 25/100mg tablet. Participants will take one tablet three times a day for the first week of the study period, increasing to two tablets three times a day for the remainder of the study period.
  Interventions: Drug: carbidopa-levodopa
- Placebo (Placebo Comparator): Participants will take one placebo tablet three times a day for the first week of the study period, increasing to two tablets three times a day for the remainder of the study period.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: carbidopa-levodopa — Motivated by the success of dopaminergic drugs in treating rigidity associated with Parkinson's disease, some neurologists have used carbidopa-levodopa to attempt to improve spasticity in ALS and PLS patients.
  Other Names: Sinemet
  Arms: carbidopa-levodopa
Drug: Placebo Oral Tablet — Placebo will be given to maintain blinding of participants and study team.
  Arms: Placebo

SUMMARY:
Motivated by the success of dopaminergic drugs in treating rigidity associated with Parkinson's disease, some neurologists have used carbidopa-levodopa (Sinemet) to attempt to improve spasticity in ALS and PLS patients. However, data on the efficacy of carbidopa/levodopa is limited. Given the limited data and potential to improve the quality of life of these patients, the effectiveness of carbidopa-levodopa in ALS and PLS patients with severe spasticity should be studied. The investigators hypothesis is that administration of carbidopa-levodopa will improve spasticity in ALS and PLS patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS or PLS
* Age greater than 18 years
* Clinically significant spasticity.

Exclusion Criteria:

* Individuals currently taking carbidopa-levodopa or with known hypersensitivity of any component of carbidopa-levodopa
* Narrow-angle glaucoma
* Current use of a non-selective monoamine oxidase inhibitor (MAOI)
* History of malignant melanoma or suspicious skin lesions
* History of depression, suicidal ideation, or psychosis
* History of myocardial infarction, ventricular arrhythmia, or severe cardiopulmonary disease
* Uncontrolled hypertension
* Asthma
* Renal disease
* Hepatic disease
* Endocrine disease
* History of peptic ulcer
* Pregnant and/or breastfeeding
* Current participation in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale - Change of spasticity severity from baseline with treatment and placebo | Weekly from screening to end of study (six weeks)
  Numerical rating scale from 0-10, where 0 is no spasticity and 10 is worst possible spasticity

SECONDARY OUTCOMES:
Visual Analog Scale - Change of pain severity from baseline with treatment and placebo | Weekly from screening to end of study (six weeks)
  Numerical rating scale from 0-10, where 0 is no pain and 10 is worst possible pain
Visual Analog Scale - Change of muscle spasm severity from baseline with treatment and placebo | Weekly from screening to end of study (six weeks)
  Numerical rating scale from 0-10, where 0 is no muscle spasm and 10 is worst possible muscle spasm
Strength | At screening, at 3 weeks (following first arm), and at 6 weeks (following second arm)
  Medical Research Council scale for muscle strength which grades power on a scale of 0 to 5 in relation to the maximum expected for that muscle, 0 being no movement observed to 5 being muscle contracts normally against full resistance.
Spasticity | At screening, at 3 weeks (following first arm), and at 6 weeks (following second arm)
  The Ashworth scale measures severity of spasticity on a scale of 1 to 5, where 1 is normal muscle tone and 5 is a rigid limb.
Upper extremity function | At screening, at 3 weeks (following first arm), and at 6 weeks (following second arm)
  9-hole peg test
Lower extremity function:10-meter Walk Test | At screening, at 3 weeks (following first arm), and at 6 weeks (following second arm)
  10-meter Walk Test is a performance measure used to assess walking speed in meters per second over a short distance.
Lower extremity function: Timed Up and Go (TUG) Test | At screening, at 3 weeks (following first arm), and at 6 weeks (following second arm)
  The TUG test measures the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down to asses a person's mobility and lower extremity function.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Miller, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT03929068/Prot_SAP_000.pdf